CLINICAL TRIAL: NCT06175728
Title: Feasibility, Usability, Acceptability and Efficacy of a Novel Leg Strengthening Device (S-Press) for Strengthening Leg Muscles and Improving Physical Impairment During Hospital Admission
Brief Title: Feasbility and Efficacy of S-Press Leg Strengthening Device
Acronym: S-PRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: NHS Northamptonshire (Unknown); JT Rehab Ltd (Industry)
Responsible Party: Principal Investigator, Tom Maden-Wilkinson, Associate Professor, Sheffield Hallam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPRESS1
Record Dates: First submitted 2023-09-06; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Deconditioning; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of S-Press (Experimental): Use of the S-Press during in patient stay alongside usual physiotherapy sessions
  Interventions: Device: S-Press

INTERVENTIONS:
Device: S-Press — Leg Strengthening Device that can be used in supine and seated positions

SUMMARY:
The proposed study will examine the use and effectiveness of a novel strength training device - The S-Press within an NHS environment. The S-Press is a portable exercise device that can be used seated or lying down and specifically targets the knee extensors and flexors. The knee extensors are particularly important in the performance of activities of daily living such as rising from a chair, walking up and down stairs and walking.

Resistance training is the most effective strategy to help to reduce muscle wasting in response to ageing or chronic disuse; however as current in-patient settings likely fail to produce an overload stimulus to the muscle for hypertrophy and strength gains, there is a need to develop new interventions and equipment to help deliver this. The S-Press is designed by a Physiotherapist with the goal of increasing muscle strength and improving physical function in patients who may be confined to their bed or chair or unable to join in with standard physiotherapy treatments.

This mixed methods study will examine the efficacy of the S-Press to improve muscle size using B-Mode Ultrasound and physical function, using sit to stand x5 with use over 6 weeks, alongside the qualitative experience of the use of the S-Press through a one to one semi structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Any in-patient admitted onto the ward sites for therapy intervention, assessed as medically stable and physically able to participate by nursing staff and able to provide informed written consent for participation.

Exclusion Criteria:

* Any patient who is unable to give informed consent.

  * Significantly confused patients - may not understand or retain the information to perform the exercises so will be excluded from this study.
  * Patients with unstable or deteriorating medical conditions or are acutely unwell with an infection.
  * Patients unable to do leg press exercise
  * Patients who have had major surgery or myocardial infarction within the past 6 months.
  * Patients who have major surgery scheduled during the intervention period.
  * Patients currently undergoing treatment for cancer
  * Patients who currently have high blood pressure that is uncontrolled (Systolic >200mmHg or Diastolic > 110mmHg)
  * Patients with a physical disability that precludes safe and adequate testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Feasbility of use of S-Press by patients | through study completion, an average of 2 weeks
  30 minute Semi Structured Interview
Feasbility of use of S-Press by Healthcare Professionals | through study completion, an average of 2 weeks
  30 minute Semi Structured Interview

SECONDARY OUTCOMES:
5x Sit to Stand time | through study completion, an average of 2 weeks
  time to complete 5 sit to stands from standardised chair
Muscle thickness | through study completion, an average of 2 weeks
  Ultrasound measurement of Vastus Lateralis
Heart rate during use | through study completion, an average of 2 weeks
  During exercise sessions
Systolic Blood Pressure during use | through study completion, an average of 2 weeks
  During exercise sessions
Diastolic Blood Pressure during use | through study completion, an average of 2 weeks
  During exercise sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Northamptonshire NHS Trust, Northampton, Northamptonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data are available on request

DOCUMENTS (1):
  • Study Protocol (2020-01-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT06175728/Prot_000.pdf